CLINICAL TRIAL: NCT04964336
Title: Decoding the B Cell Response in Multiple Sclerosis
Brief Title: An Observational Study to Investigate the Role of B Cells in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Andreas Lossius, Associate Professor, University of Oslo
Other Study IDs: 314376 - FORSKER20
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis: Patients with relapsing-remitting multiple sclerosis
  Interventions: Other: Analysis of B cells

INTERVENTIONS:
Other: Analysis of B cells — B cells from blood and cerebrospinal fluid will be analyzed using RNA-seq

SUMMARY:
Multiple sclerosis (MS) typically afflict young people in their twenties, when they start a career and establish a family. The disease thus imposes a severe impact on quality of life and heavy economic burdens on society. Critical barriers to progress in the field are the lack of knowledge of relevant immune cell subsets driving the pathology and the targets of the immune response within the central nervous system. In this project, we will test the hypothesis that a subgroup of MS patients is defined by a genetically determined B cell response against specific antigenic epitopes. The hypothesis is based on our recent, pioneering results showing that approximately half of MS patients have a restricted population of B cells in the cerebrospinal fluid defined by polymorphisms in the constant heavy-chain of the immunoglobulin B cell receptor, the G1m1 allotype. Here, we aim to characterize the G1m1 B cells, to disentangle the genetic basis of the B cell response, and to identify the molecular targets.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and brain MRI scans strongly suggestive of multiple sclerosis according to the 2017 McDonald revisions
* Intrathecal immunoglobulin G synthesis
* Age > 18 years

Exclusion Criteria:

* Treatment with immunomodulatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under diagnostic work-up for multiple sclerosis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The transcriptome of B cells from blood and cerebrospinal fluid | 1 day (subject inclusion)
The immunglobulin receptors of B cells from blood and cerebrospinal fluid | 1 day (subject inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Lossius, Principal Investigator — University of Oslo
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No